#### **CONSENT FOR RESEARCH**

The Pennsylvania State University

Title of Project: Smart Parents – Safe and Healthy Kids

Principal Investigator: Kate Guastaferro, Ph.D.

Address: 418 Health & Human Development Building, University Park, PA 16802
Telephone Number: (814) 863-9795
Email Address: kmg55@psu.edu

Subject's Printed Name:

We are asking you to be in a research study. This form gives you information about the research.

Whether or not you take part is up to you. You can choose not to take part. You can agree to take part and later change your mind. Your decision will not be held against you.

Please ask questions about anything that is unclear to you and take your time to make your choice.

# 1. Why is this research study being done?

We are asking you to be in this research because you have signed up for Parents as Teachers. This research is being done to better understand ways in which we can support parents in improving their children's health and well-being by evaluating the potential benefit of additional program content in improving parents' knowledge and skills. Approximately 124 people will take part in this research study nationwide.

# 2. What will happen in this research study?

As you participate in the Parents as Teachers program, we will ask you to complete a brief survey at four time points, including today. After you complete 5 foundational PAT visits, we will ask you to participate in an extra session to learn additional material about children's healthy sexual development, how to talk to your child about sexual abuse, and skills to keep your child safe.

The surveys include questions about your behavior, your child's behavior, your and your child's relationship, your attitudes and opinions about parenting, and your thoughts on how the extra session was delivered to you. Some of the questions are personal in nature and address sensitive topics, including alcohol/drug use, emotional problems, potentially illegal behaviors, and recognizing/preventing child maltreatment. You are free to skip any questions that you would prefer not to answer, and your answers will be kept confidential.

Some subjects will be asked to allow their last session to be audio recorded. The purpose of the audio recording is not to review what your responses were, but simply to confirm that the provider presented all of the program information. You are free to skip the audio recording if you do not want to participate in that part.

If you choose not to participate in the research, you would not complete the surveys and you would not have the extra session.

# 3. What are the risks and possible discomforts from being in this research study?

You may find some of the program content upsetting or uncomfortable to talk about. These risks are not more than you might experience in everyday life as a parent, but your provider is experienced in discussing these topics and available to help should you need it. Some of the survey questions are personal in nature and cover sensitive topics or might cause discomfort. You do not have to answer any questions you do not want to, and your answers will be kept confidential. If you participate in the audio recording, you may ask your provider to turn off the device at any time. This way if you wish to discuss a sensitive topic it is not recorded.

There is a risk of loss of confidentiality if your information or your identity is obtained by someone other than the investigators, but precautions will be taken to prevent this from happening. The confidentiality of your data created by you or by the researchers will be maintained to the degree permitted by the technology used. Absolute confidentiality cannot be guaranteed.

# 4. What are the possible benefits from being in this research study?

# 4a. What are the possible benefits to you?

By participating in this research, you will learn skills to help keep your child safe from victimization.

# 4b. What are the possible benefits to others?

Families who become engaged with agencies, such as Child and Youth Services, will benefit from your participation in this study. Your insight will help us create programs that best meet the needs of children and parents.

# 5. What other options are available instead of being in this research study?

You may decide not to participate in the surveys. Your decision not to participate will not affect your ability to complete Parents as Teachers.

# 6. How long will you take part in this research study?

Your total participation in the program will last at least 6 weeks. Your total participation in the surveys will take about an hour (the first survey will take about 25 minutes, the second survey about 10 minutes, the third survey about 15 minutes, and the last survey about 10 minutes).

# 7. How will your privacy and confidentiality be protected if you decide to take part in this research study?

Efforts will be made to limit the use and sharing of your personal research information to people who have a need to review this information. Your research records will be labeled with a unique code number and kept in a locked filing cabinet and in a password-protected file on a secure server. An electronic list that matches your name with your code number will be kept in a separate password-protected file on a secure server at our office. In the event of any publication or presentation resulting from the research, no personally identifiable information will be shared.

If you participate in the audio recording portion, recordings will be labeled with the provider's code number and secured in a password-protected file on a secure server. Only study team members will have access to these recordings and they will be destroyed three years after the study is closed.

We will do our best to keep your participation in this research study confidential to the extent permitted by law. However, it is possible that other people may find out about your participation in this research study. For example, the following people/groups may check and copy records about this research.

- The Office for Human Research Protections in the U. S. Department of Health and Human Services
- The Institutional Review Board (a committee that reviews and approves research studies) and
- The Office for Research Protections.

Some of these records could contain information that personally identifies you.

Reasonable efforts will be made to keep the personal information in your research record private. However, absolute confidentiality cannot be guaranteed. The research team is required by law to report information about suspected child abuse to appropriate authorities.

## 8. Will you be paid or receive credit to take part in this research study?

You will be compensated for completing each of the three surveys:

- \$10 for the first survey today
- \$10 for the second survey about five weeks later

- \$10 for the third survey one week later after the additional program module
- \$20 for the final survey one month later

# 9. What are your rights if you take part in this research study?

Taking part in this research study is voluntary.

- You do not have to be in this research.
- If you choose to be in this research, you have the right to stop at any time.
- If you decide not to be in this research or if you decide to stop at a later date, there will be no penalty or loss of benefits to which you are entitled.

# 10. If you have questions or concerns about this research study, whom should you call?

Please call the head of the research study, Dr. Kate Guastaferro, at (814) 863-9795 if you:

- Have questions, complaints or concerns about the research.
- Believe you may have been harmed by being in the research study.

You may also contact the Office for Research Protections at (814) 865-1775, ORProtections@psu.edu if you:

- Have questions regarding your rights as a person in a research study.
- Have concerns or general questions about the research.
- Cannot reach the research team or wish to offer input or to talk to someone else about any concerns related to the research.

Your signature below means that you have explained the research to the subject or subject representative and

# **INFORMED CONSENT TO TAKE PART IN RESEARCH**

# **Signature of Person Obtaining Informed Consent**

| have answered any questions he/she has about the research. | | |
|---|---|---|
| Signature of person who explained this res<br>(Only approved investigators for this resea | | Printed Name research and obtain informed consent.) |
| Signature of Person Giving Informed Consent Before making the decision about being in this research you should have: • Discussed this research study with an investigator, • Read the information in this form, and • Had the opportunity to ask any questions you may have. Your signature below means that you have received this information, have asked the questions you currently have about the research and those questions have been answered. You will receive a copy of the signed and dated form to keep for future reference. By signing this consent form, you indicate that you voluntarily choose to be in this research and agree to allow your information to be used and shared as described above. | | |
| Signature of Subject | Date | Printed Name |

#### CONSENT FOR RESEARCH

The Pennsylvania State University

Title of Project: Smart Parents – Safe and Healthy Kids

Principal Investigator: Kate Guastaferro, Ph.D.

Address: 418 Health & Human Development Building, University Park, PA 16802 Telephone Number: (814) 863-9795 Email Address: <a href="mailto:kmg55@psu.edu">kmg55@psu.edu</a>

| Subject's Printed Name: |
|-------------------------|

We are asking you to be in a research study. This form gives you information about the research.

Whether or not you take part is up to you. You can choose not to take part. You can agree to take part and later change your mind. Your decision will not be held against you.

Please ask questions about anything that is unclear to you and take your time to make your choice.

# 1. Why is this research study being done?

We are asking you to be in this research because you have signed up for Parents as Teachers. This research is being done to better understand ways in which we can support parents in improving their children's health and well-being by evaluating the potential benefit of additional program content in improving parents' knowledge and skills. Approximately 124 people will take part in this research study nationwide.

# 2. What will happen in this research study?

As you participate in the Parents as Teachers program, we will ask you to complete a brief survey at four time points, including today.

The surveys include questions about your behavior, your child's behavior, your and your child's relationship, and your attitudes and opinions about parenting. Some of the questions are personal in nature and address sensitive topics, including alcohol/drug use, emotional problems, potentially illegal behaviors, and recognizing/preventing child maltreatment. You are free to skip any questions that you would prefer not to answer, and your answers will be kept confidential.

If you choose not to participate in the research, you would not complete the surveys.

# 3. What are the risks and possible discomforts from being in this research study?

Some of the survey questions are personal in nature and cover sensitive topics or might cause discomfort. You do not have to answer any questions you do not want to, and your answers will be kept confidential.

There is a risk of loss of confidentiality if your information or your identity is obtained by someone other than the investigators, but precautions will be taken to prevent this from happening. The confidentiality of your data created by you or by the researchers will be maintained to the degree permitted by the technology used. Absolute confidentiality cannot be guaranteed.

## 4. What are the possible benefits from your participation in this research study?

Families who become engaged with agencies, such as Child and Youth Services, will benefit from your participation in this study. Your insight will help us create programs that best meet the needs of children and parents.

# 5. What other options are available instead of being in this research study?

You may decide not to participate in the research. Your decision not to participate will not affect your ability to complete Parents as Teachers.

# 6. How long will you take part in this research study?

Your total participation in the foundational portion of the program will last at least 5 weeks. Your total participation in the surveys will take about 55 minutes (the first survey will take about 25 minutes, and the other three times we ask you to complete a survey, it will take you about 10 minutes each).

# 7. How will your privacy and confidentiality be protected if you decide to take part in this research study?

Efforts will be made to limit the use and sharing of your personal research information to people who have a need to review this information. Your research records will be labeled with a unique code number and kept in a locked filing cabinet and in a password-protected file on a secure server. An electronic list that matches your name with your code number will be kept in a separate password-protected file on a secure server at our office. In the event of any publication or presentation resulting from the research, no personally identifiable information will be shared.

We will do our best to keep your participation in this research study confidential to the extent permitted by law. However, it is possible that other people may find out about your participation in this research study. For example, the following people/groups may check and copy records about this research.

- The Office for Human Research Protections in the U. S. Department of Health and Human Services
- The Institutional Review Board (a committee that reviews and approves research studies) and
- The Office for Research Protections.

Some of these records could contain information that personally identifies you.

Reasonable efforts will be made to keep the personal information in your research record private. However, absolute confidentiality cannot be guaranteed. The research team is required by law to report information about suspected child abuse to appropriate authorities.

#### 8. Will you be paid or receive credit to take part in this research study?

You will be compensated for completing each of the four surveys:

- \$10 for the first survey today
- \$10 for the second survey about 5 weeks later
- \$10 for the third survey one week later
- \$20 for the third survey one month later

# 9. What are your rights if you take part in this research study?

Taking part in this research study is voluntary.

- You do not have to be in this research.
- If you choose to be in this research, you have the right to stop at any time.
- If you decide not to be in this research or if you decide to stop at a later date, there will be no penalty or loss of benefits to which you are entitled.

## 10. If you have questions or concerns about this research study, whom should you call?

Please call the head of the research study, Dr. Kate Guastaferro, at (814) 863-9795 if you:

- Have questions, complaints or concerns about the research.
- Believe you may have been harmed by being in the research study.

You may also contact the Office for Research Protections at (814) 865-1775, ORProtections@psu.edu if you:

- Have questions regarding your rights as a person in a research study.
- Have concerns or general questions about the research.
- Cannot reach the research team or wish to offer input or to talk to someone else about any concerns related to the research.

# **INFORMED CONSENT TO TAKE PART IN RESEARCH**

# **Signature of Person Obtaining Informed Consent**

| Your signature below means that your representative and have answered | • | • |
|---|---|---|
| Signature of person who explained t (Only approved investigators for this | | Printed Name esearch and obtain informed consent.) |
| | eing in this research you sho<br>y with an investigator,<br>form, and<br>any questions you may have<br>u have received this informa<br>questions have been answer | |
| By signing this consent form, you indallow your information to be used an | | noose to be in this research and agree to<br>re. |
| Signature of Subject | <br>Date | Printed Name |